CLINICAL TRIAL: NCT02793544
Title: A Multi-Center, Phase II Trial of HLA-Mismatched Unrelated Donor Bone Marrow Transplantation With Post-Transplantation Cyclophosphamide for Patients With Hematologic Malignancies
Brief Title: HLA-Mismatched Unrelated Donor Bone Marrow Transplantation With Post-Transplantation Cyclophosphamide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-MMUD
Record Dates: First submitted 2016-05-31; First posted 2016-06-08 (Estimated); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Myelodysplastic Syndrome (MDS); Chronic Lymphocytic Leukemia (CLL); Chemotherapy-sensitive Lymphoma; Acute Lymphoblastic Leukemia (ALL)/T Lymphoblastic Lymphoma; Acute Myelogenous Leukemia (AML); Acute Biphenotypic Leukemia (ABL); Acute Undifferentiated Leukemia (AUL)
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Lymphocytic, Chronic, B-Cell; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation; Busulfan; Sirolimus; Mycophenolic Acid; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Regimen A (RIC: Flu/Cy/TBI) (Active Comparator): 1. Fludarabine 30 mg/m2/day IV on Days -6, -5, -4, -3, -2
  2. Cyclophosphamide 14.5 mg/kg/day IV on Days -6, -5
  3. Total Body Irradiation (TBI) 200cGy on Day -1
  4. Infusion of non-T-cell depleted bone marrow on Day 0
  Although a schedule is proposed above, the regimen can be given according to institutional standards as long as the prescribed doses are the same as in the recommended regimen above.
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide 14.5 mg/kg/day IV on Days -6, -5; Radiation: Total Body Irradiation (TBI) 200cGy on Day -1; Procedure: Infusion of non-T-cell depleted bone marrow on Day 0; Drug: Post-HCT Cyclophosphamide 50mg/kg IV on Day+3, +4; Drug: Sirolimus; Drug: Mycophenolate mofetil; Drug: G-CSF; Drug: Pre-HCT Mesna on Days -6 and -5; Drug: Post-HCT Mesna
- Regimen B 2a (FIC: Bu/Cy) (Active Comparator): 1. Busulfan ≥ 9mg/kg total dose on Days -6, -5, -4, -3 (IV or PO)
  2. Cyclophosphamide 50mg/kg/day IV on Days -2,-1
  3. Infusion of non-T-cell depleted bone marrow on Day 0
  Although a schedule is proposed above, the regimen can be given according to institutional standards as long as the prescribed doses are the same as in the recommended regimen above.
  Interventions: Procedure: Infusion of non-T-cell depleted bone marrow on Day 0; Drug: Busulfan; Drug: Cyclophosphamide 50mg/kg/day IV on Days -2,-1; Drug: Post-HCT Cyclophosphamide 50mg/kg IV on Day+3, +4; Drug: Sirolimus; Drug: Mycophenolate mofetil; Drug: G-CSF; Drug: Pre-HCT Mesna on Days -2 and -1; Drug: Post-HCT Mesna
- Regimen B 2b (FIC: Bu/Flu) (Active Comparator): 1. Busulfan ≥ 9mg/kg total dose on Days -6, -5, -4, -3 (IV or PO)
  2. Fludarabine 30 mg/m2/day IV on Days -6, -5, -4, -3, -2
  3. Infusion of non-T-cell depleted bone marrow on Day 0
  Although a schedule is proposed above, the regimen can be given according to institutional standards as long as the prescribed doses are the same as in the recommended regimen above.
  Interventions: Drug: Fludarabine; Procedure: Infusion of non-T-cell depleted bone marrow on Day 0; Drug: Busulfan; Drug: Post-HCT Cyclophosphamide 50mg/kg IV on Day+3, +4; Drug: Sirolimus; Drug: Mycophenolate mofetil; Drug: G-CSF; Drug: Post-HCT Mesna
- Regimen C (FIC: Cy/TBI) (Active Comparator): 1. Cyclophosphamide 50mg/kg/day IV on Days -5,-4
  2. Total Body Irradiation (TBI) 200cGy twice a day on Days -3, -2, -1
  3. Infusion of non-T-cell depleted bone marrow on Day 0
  Although a schedule is proposed above, the regimen can be given according to institutional standards as long as the prescribed doses are the same as in the recommended regimen above.
  Interventions: Procedure: Infusion of non-T-cell depleted bone marrow on Day 0; Drug: Cyclophosphamide 50mg/kg/day IV on Days -5,-4; Radiation: Total Body Irradiation (TBI) 200cGy twice a day on Days -3, -2, -1; Drug: Post-HCT Cyclophosphamide 50mg/kg IV on Day+3, +4; Drug: Sirolimus; Drug: Mycophenolate mofetil; Drug: G-CSF; Drug: Pre-HCT Mesna on Days -5 and -4; Drug: Post-HCT Mesna

INTERVENTIONS:
Drug: Fludarabine — * Fludarabine 30 mg/m2/day (adjusted for renal function) is administered over a 30-60 minute IV infusion on Days -6 through -2 (maximum cumulative dose, 150 mg/m2).
  * The body surface area (BSA) for fludarabine dosing is based on adjusted ideal body weight (IBW) (Appendix K).
  * creatinine clearance may change during the days fludarabine is given. Adjustment in fludarabine dose due to creatinine changes during conditioning is permitted.
  Other Names: Fludara®
  Arms: Regimen A (RIC: Flu/Cy/TBI); Regimen B 2b (FIC: Bu/Flu)
Drug: Cyclophosphamide 14.5 mg/kg/day IV on Days -6, -5 — * Cy 14.5 mg/kg/day is administered as a 1-2 hour IV infusion on Days -6 and -5 after hydration.
  * Use of Mesna and dosing will be done according to institutional standards. A recommended approach is as follows: Mesna IV dose of ≥ 80% of the total daily dose of Cy and given in divided doses 30 minutes before and at 3, 6, and 8-9 hours after completion of Cy.
  * Hydration prior to Cy may be given according to institutional guideline.
  * Cy and mesna are dosed according to adjusted IBW (Appendix K), unless the subject weighs less than IBW, in which case these drugs will be dosed according to actual weight.
  Other Names: Cytoxan®
  Arms: Regimen A (RIC: Flu/Cy/TBI)
Radiation: Total Body Irradiation (TBI) 200cGy on Day -1 — * 200 cGy TBI is administered in a single fraction on Day -1.
  * Radiation sources, dose rates, and shielding follow institutional practice.
  Arms: Regimen A (RIC: Flu/Cy/TBI)
Procedure: Infusion of non-T-cell depleted bone marrow on Day 0 — * On Day 0, the harvested bone marrow is infused.
  * Donor bone marrow will be harvested with a target yield of 4 x 108 nucleated cells/kg recipient weight.
  * The lowest acceptable nucleated cells yield is 1.5 x 108 cells/kg recipient weight.
Drug: Busulfan — * Busulfan ≥ 9mg/kg total dose (IV or PO) on Days -6, -5, -4, -3 (PK monitoring required to achieve a daily area under the curve (AUC) target of 4800-5300 μM*min (Perkins et al., 2012))
  * Busulfan dosing is based on adjusted IBW (Appendix K)
  Other Names: Busulfex®
  Arms: Regimen B 2a (FIC: Bu/Cy); Regimen B 2b (FIC: Bu/Flu)
Drug: Cyclophosphamide 50mg/kg/day IV on Days -2,-1 — * Cy 50mg/kg/day is administered as a 1-2 hour IV infusion on Days -2 and -1 after hydration.
  * Use of Mesna and dosing will be done according to institutional standards. A recommended approach is as follows: Mesna IV dose of ≥ 80% of the total daily dose of Cy and given in divided doses 30 minutes before and at 3, 6, and 8-9 hours after completion of Cy.
  * Hydration prior to Cy may be given according to institutional guideline.
  * Cy and mesna are dosed according to adjusted IBW (Appendix K), unless the subject weighs less than IBW, in which case these drugs will be dosed according to actual weight.
  Other Names: Cytoxan®
  Arms: Regimen B 2a (FIC: Bu/Cy)
Drug: Cyclophosphamide 50mg/kg/day IV on Days -5,-4 — * Cy 50mg/kg/day is administered as a 1-2 hour IV infusion on Days -5 and -4 after hydration.
  * Use of Mesna and dosing will be done according to institutional standards. A recommended approach is as follows: Mesna IV dose of ≥ 80% of the total daily dose of Cy and given in divided doses 30 minutes before and at 3, 6, and 8-9 hours after completion of Cy.
  * Hydration prior to Cy may be given according to institutional guideline.
  * Cy and mesna are dosed according to adjusted IBW (Appendix K), unless the subject weighs less than IBW, in which case these drugs will be dosed according to actual weight.
  Other Names: Cytoxan®
  Arms: Regimen C (FIC: Cy/TBI)
Radiation: Total Body Irradiation (TBI) 200cGy twice a day on Days -3, -2, -1 — * 200cGy TBI is administered in twice daily on Days -3, -2, and -1.
  * Radiation sources, dose rates, and shielding follow institutional practice.
  Arms: Regimen C (FIC: Cy/TBI)
Drug: Post-HCT Cyclophosphamide 50mg/kg IV on Day+3, +4 — * Cy 50mg/kg IV, over 1-2 hours (depending on volume), is given on Day+3 (ideally between 60 and 72 hours after bone marrow infusion) and on Day+4 (approximately 24 hours after Day+3 Cy).
  * Hydration with Cy, management of volume status, and monitoring for hemorrhagic cystitis will follow institutional standards.
  * Mesna is required. Mesna IV dose must be ≥ 80% of the total daily dose of Cy and given in divided doses 30 minutes before and at 3, 6, and 8-9 hours after completion of Cy.
  * Cy is dosed according to IBW, unless the subject weighs less than IBW, in which case these drugs will be dosed according to actual body weight.
Drug: Sirolimus — * Sirolimus dosing is based on adjusted IBW (Appendix K).
  * Sirolimus prophylaxis is discontinued after the last dose on Day+180, or may be continued if there is GVHD.
  For subjects ≥ 18 years old:
  * A one-time sirolimus loading dose, 6 mg PO, is given on Day+5, at least 24 hours after Cy completion.
  * Sirolimus is then continued at a maintenance dose (starting dose 2 mg PO QD), with dose adjustments to maintain a trough of 5 - 15 ng/mL as measured by high performance liquid chromatography (HPLC) or immunoassay.
  For subjects < 18 years old:
  * A one-time sirolimus loading dose, 3 mg/m2 PO with the dose not to exceed 6 mg, is given on Day+5, at least 24 hours after Cy completion.
  * Sirolimus is then continued at a maintenance dose (starting dose 1 mg/m2 PO QD, maximum 2 mg PO QD), with dose adjustments to maintain a trough of 5 - 15 ng/mL as measured by HPLC or immunoassay.
  Other Names: rapamycin; Rapamune®
Drug: Mycophenolate mofetil — MMF begins on Day+5, at least 24 hours after completion of PTCy. MMF dose is 15 mg/kg PO TID (adjusted IBW (Appendix K)) with total daily dose not to exceed 3 grams (i.e. maximum 1 g PO TID).
  An equivalent IV dose (1:1 conversion) may instead be given. MMF prophylaxis is discontinued after the last dose on Day+35, or may be continued if there is GVHD.
  Other Names: MMF; Cellcept®
Drug: G-CSF — Granulocyte-colony stimulating factor (G-CSF): filgrastim or a biosimilar begins on Day+5 at a dose of 5 mcg/kg/day (actual body weight) IV or subcutaneously (SC) (rounding to the nearest vial dose is allowed), until the absolute neutrophil count (ANC) is ≥ 1,000/mm3 over the course of 3 consecutive days.
  Additional G-CSF may be administered as warranted.
  Other Names: filgrastim
Drug: Pre-HCT Mesna on Days -6 and -5 — Use of Mesna and dosing will be done according to institutional standards. A recommended approach is as follows: Mesna IV dose of ≥ 80% of the total daily dose of Cy and given in divided doses 30 minutes before and at 3, 6, and 8-9 hours after completion of Cy.
  Mesna is dosed according to adjusted IBW (Appendix K), unless the subject weighs less than IBW, in which case Mesna will be dosed according to actual weight.
  Arms: Regimen A (RIC: Flu/Cy/TBI)
Drug: Pre-HCT Mesna on Days -2 and -1 — Use of Mesna and dosing will be done according to institutional standards. A recommended approach is as follows: Mesna IV dose of ≥ 80% of the total daily dose of Cy and given in divided doses 30 minutes before and at 3, 6, and 8-9 hours after completion of Cy.
  Mesna is dosed according to adjusted IBW (Appendix K), unless the subject weighs less than IBW, in which case Mesna will be dosed according to actual weight.
  Arms: Regimen B 2a (FIC: Bu/Cy)
Drug: Pre-HCT Mesna on Days -5 and -4 — Use of Mesna and dosing will be done according to institutional standards. A recommended approach is as follows: Mesna IV dose of ≥ 80% of the total daily dose of Cy and given in divided doses 30 minutes before and at 3, 6, and 8-9 hours after completion of Cy.
  Mesna is dosed according to adjusted IBW (Appendix K), unless the subject weighs less than IBW, in which case Mesna will be dosed according to actual weight.
  Arms: Regimen C (FIC: Cy/TBI)
Drug: Post-HCT Mesna — Mesna is required. Mesna IV dose must be ≥ 80% of the total daily dose of Cy and given in divided doses 30 minutes before and at 3, 6, and 8-9 hours after completion of Cy on Day+3 and Day+4.
  Mesna is dosed according to IBW, unless the subject weighs less than IBW, in which case Mesna will be dosed according to actual body weight.

SUMMARY:
This is a multi-center, single arm Phase II study of hematopoietic cell transplantation (HCT) using human leukocyte antigen (HLA)-mismatched unrelated bone marrow transplantation donors and post-transplantation cyclophosphamide (PTCy), sirolimus and mycophenolate mofetil (MMF) for graft versus host disease (GVHD) prophylaxis in patients with hematologic malignancies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 15 years and < 71 years at the time of signing the informed consent form
2. Partially HLA-mismatched unrelated donor: HLA typing will be performed at high resolution (allele level) for the HLA-A, -B, -C, and -DRB1 loci; a minimum match of 4/8 at HLA-A, -B, -C, and -DRB1 is required
3. Product planned for infusion is bone marrow
4. Disease and disease status:

   1. Acute Leukemias or T lymphoblastic lymphoma in 1st or subsequent complete remission (CR): Acute lymphoblastic leukemia (ALL)/T lymphoblastic lymphoma; acute myelogenous leukemia (AML); acute biphenotypic leukemia (ABL); acute undifferentiated leukemia (AUL)
   2. Myelodysplastic Syndrome (MDS), fulfilling the following criteria: Subjects with de novo MDS who have or have previously had Intermediate-2 or High risk disease as determined by the International Prognostic Scoring System (IPSS). Current Intermediate-2 or High risk disease is not a requirement; Subjects must have < 20% bone marrow blasts, assessed within 60 days of informed consent; Subjects may have received prior therapy for the treatment of MDS prior to enrollment
   3. Chronic Lymphocytic Leukemia (CLL) in CR if RIC is to be used; in CR or partial response (PR) if FIC is to be used
   4. Chronic myeloid leukemia (CML) in 1st or subsequent chronic phase characterized by <10% blasts in the blood or bone marrow.
   5. Chemotherapy-sensitive lymphoma in status other than 1st CR
5. Performance status: Karnofsky or Lansky score ≥ 60% (Appendix A)
6. Adequate organ function defined as:

   1. Cardiac: left ventricular ejection fraction (LVEF) at rest ≥ 35% (RIC cohort) or LVEF at rest ≥ 40% (FIC cohort), or left ventricular shortening fraction (LVFS) ≥ 25%
   2. Pulmonary: diffusing capacity of the lungs for carbon monoxide (DLCO), forced expiratory volume (FEV1), forced vital capacity (FVC) ≥ 50% predicted by pulmonary function tests (PFTs)
   3. Hepatic: total bilirubin ≤ 2.5 mg/dL, and alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase (ALP) < 5 x upper limit of (ULN) (unless disease related)
   4. Renal: serum creatinine (SCr) within normal range for age (see table 2.3). If SCr is outside normal range for age, creatinine clearance (CrCl) > 40 mL/min/1.73m2 must be obtained (measured by 24-hour (hr) urine specimen or nuclear glomerular filtration rate (GFR), or calculated GFR (by Cockcroft-Gault formula for those aged ≥ 18 years; by Original Schwartz estimate for those < 18 years))
7. Subjects ≥ 18 years of age must have the ability to give informed consent according to applicable regulatory and local institutional requirements. Legal guardian permission must be obtained for subjects < 18 years of age. Pediatric subjects will be included in age appropriate discussion in order to obtain assent.
8. Subjects with documentation of confirmed HIV-1 infection (i.e. HIV-positive), and a hematologic malignancy who meets all other eligibility requirements must:

   1. Receive only RIC regimen (i.e. Regimen A)
   2. Be willing to comply with effective antiretroviral therapy (ARV)
   3. Have achieved a sustained virologic response for 12 weeks after cessation of hepatitis C antiviral treatment (in HIV-positive subjects with hepatitis C)

Exclusion Criteria:

1. HLA-matched related or 8/8 allele matched (HLA-A, -B, -C, -DRB1) unrelated donor available. This exclusion does not apply to HIV-positive subjects who have a CCR5delta32 homozygous donor.
2. Autologous HCT < 3 months prior to the time of signing the informed consent form
3. Females who are breast-feeding or pregnant
4. HIV-positive subjects:

   1. Acquired immunodeficiency syndrome (AIDS) related syndromes or symptoms that may pose an excessive risk for transplantation-related morbidity as determined by the Treatment Review Committee (see Appendix D).
   2. Untreatable HIV infection due to multidrug ARV resistance. Subjects with a detectable or standard viral load > 750 copies/mL should be evaluated with an HIV drug resistance test (HIV-1 genotype). The results should be included as part of the ARV review (described in Appendix D).
   3. May not be currently prescribed ritonavir, cobacistat and/or zidovudine
5. Current uncontrolled bacterial, viral or fungal infection (currently taking medication with evidence of progression of clinical symptoms or radiologic findings)
6. Prior allogeneic HCT
7. History of primary idiopathic myelofibrosis
8. MDS subjects may not receive RIC and must be < 50 years of age at the time of signing the informed consent form

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Bolaños Meade, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Centre at Johns Hopkins; Bronwen E. Shaw, MD, PhD, Study Chair — CIBMTR/Medical College of Wisconsin
Locations (11):
- United States (11):
  - Shands HealthCare & University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Maryland Greenebaum Cancer Center, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Cancer Center - Adults, New York, New York
  - University of North Carolina Hospitals, Chapel Hill, North Carolina
  - Ohio State Medical Center, James Cancer Center, Columbus, Ohio
  - Virginia Commonwealth University Massey Cancer Center Bone Marrow Transplant Program, Richmond, Virginia
  - Froedtert Memorial Lutheran Hospital, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Shaw BE, Jimenez-Jimenez AM, Burns LJ, Logan BR, Khimani F, Shaffer BC, Shah NN, Mussetter A, Tang XY, McCarty JM, Alavi A, Farhadfar N, Jamieson K, Hardy NM, Choe H, Ambinder RF, Anasetti C, Perales MA, Spellman SR, Howard A, Komanduri KV, Luznik L, Norkin M, Pidala JA, Ratanatharathorn V, Confer DL, Devine SM, Horowitz MM, Bolanos-Meade J. National Marrow Donor Program-Sponsored Multicenter, Phase II Trial of HLA-Mismatched Unrelated Donor Bone Marrow Transplantation Using Post-Transplant Cyclophosphamide. J Clin Oncol. 2021 Jun 20;39(18):1971-1982. doi: 10.1200/JCO.20.03502. Epub 2021 Apr 27. PMID 33905264

RESULTS

PARTICIPANT FLOW:
Groups:
- Myeloablative Conditioning (MAC): Participants received one of three regimens: cyclophosphamide and total body irradiation; busulfan and cyclophosphamide; or fludarabine and busulfan
- Reduced Intensity Conditioning (RIC): Participants received one of two regimens: fludarabine, cyclophosphamide, and low-dose total body irradiation
Period: Overall Study
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Started | 40 | 40
Completed | 27 | 32
Not Completed | 13 | 8
Not completed — Death | 10 | 8
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC) | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Median (Full Range); unit: years] | 48.5 [18 to 66] | 59.5 [23 to 70] | 51.5 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 21 | 38
  Male | 23 | 19 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 7 | 19
  Not Hispanic or Latino | 28 | 33 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 6 | 15
  White | 29 | 31 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 40 | 80
Karnofsky/Lansky performance score [Count of Participants; unit: Participants] — Performance score (Karnofsky if ≥ 16 years, Lansky score if < 16 years) of participants at baseline. The range is 0 to 100 with 100 being the best.
  Participants
    70 | 2 | 1 | 3
    80 | 12 | 12 | 24
    90 | 21 | 17 | 38
    100 | 5 | 10 | 15
HCT Comorbidity Index score [Count of Participants; unit: Participants] — Hematopoietic Cell Transplantation Comorbidity Index (HCT-CI) is a tool to assess the risk of non-relapse (NRM) mortality and survival. Scores are divided into 3 groups according to risk: low risk (0), intermediate risk (1-2), and high risk (≥ 3). A higher score indicates higher risk of NRM and overall mortality.
  Participants
    0 | 4 | 9 | 13
    1 | 2 | 8 | 10
    2 | 10 | 4 | 14
    3+ | 24 | 19 | 43
Primary Disease [Count of Participants; unit: Participants]
  Acute leukemia | 37 | 23 | 60
  MDS | 2 | 0 | 2
  CLL | 0 | 3 | 3
  Lymphoma | 1 | 14 | 15
Disease status pre-HCT [Count of Participants; unit: Participants]
  CR1 | 32 | 23 | 55
  CR2+ | 6 | 6 | 12
  CR | 1 | 3 | 4
  Progression/Relapse | 0 | 3 | 3
  PIF | 0 | 5 | 5
  HI | 1 | 0 | 1
Refined disease risk index [Count of Participants; unit: Participants] — Disease risk index is categorized based on disease, stage, cytogenetics for AML, ALL, CML, CLL, MDS, MPN, HL, NHL and PCD.
  Participants
    Low | 3 | 6 | 9
    Intermediate | 29 | 21 | 50
    High | 3 | 7 | 10
    Very high | 0 | 3 | 3
    N/A | 5 | 3 | 8
CMV serostatus [Count of Participants; unit: Participants]
  Negative | 16 | 18 | 34
  Positive | 24 | 22 | 46
Conditioning Regimen [Count of Participants; unit: Participants]
  TBI and Cy | 6 | 0 | 6
  TBI, CY, and Flu | 0 | 40 | 40
  Bu and Cy | 3 | 0 | 3
  Bu and Flu | 31 | 0 | 31
HLA match, categorical [Count of Participants; unit: Participants]
  7/8 | 26 | 23 | 49
  6/8 | 8 | 11 | 19
  5/8 | 5 | 2 | 7
  4/8 | 1 | 4 | 5
Infused total nucleated cells x10^8/kg [Median (Full Range); unit: cells x10^8/kg] | 2.81 [0.6 to 520.8] | 2.8 [0.76 to 5.8] | 2.8 [0.6 to 520.8]
Infused CD34 cells, x10^6/kg [Median (Full Range); unit: cells x10^6/kg] | 2.72 [0.89 to 5.24] | 2.2 [0.39 to 6.23] | 2.66 [0.39 to 6.23]
Donor age [Count of Participants; unit: Participants]
  18-29 years of age | 24 | 23 | 47
  30-39 years of age | 9 | 11 | 20
  40-49 years of age | 4 | 6 | 10
  50-59 years of age | 3 | 0 | 3
Donor Sex [Count of Participants; unit: Participants]
  Male | 20 | 24 | 44
  Female | 20 | 16 | 36
Donor/recipient sex [Count of Participants; unit: Participants]
  M-M | 12 | 12 | 24
  M-F | 8 | 12 | 20
  F-M | 11 | 7 | 18
  F-F | 9 | 9 | 18
Donor/recipient CMV serostatus [Count of Participants; unit: Participants]
  +/+ | 18 | 13 | 31
  +/- | 6 | 5 | 11
  -/+ | 9 | 10 | 19
  -/- | 7 | 12 | 19
Donor/recipient ABO match [Count of Participants; unit: Participants]
  Matched | 20 | 24 | 44
  Minor mismatch | 12 | 5 | 17
  Major mismatch | 8 | 8 | 16
  Bi-directional | 0 | 3 | 3
HIV infection pre-HCT [Count of Participants; unit: Participants]
  No | 40 | 36 | 76
  Yes | 0 | 4 | 4
Disease and disease status at HCT [Count of Participants; unit: Participants]
  AML (CR1) | 22 | 10 | 32
  AML (CR2+) | 1 | 2 | 3
  AML (PIF) | 0 | 2 | 2
  ALL (CR1) | 7 | 6 | 13
  ALL (CR2+) | 3 | 1 | 4
  CLL (CR) | 0 | 3 | 3
  MDS (CR) | 1 | 0 | 1
  MDS (HI) | 1 | 0 | 1
  Other acute leukemia (CR1) | 3 | 0 | 3
  Other acute leukemia (CR2+) | 1 | 0 | 1
  NHL (CR1) | 0 | 5 | 5
  NHL (CR2+) | 1 | 3 | 4
  NHL (Relapse) | 0 | 2 | 2
  NHL (PIF) | 0 | 1 | 1
  HL (CR1) | 0 | 2 | 2
  HL (Relapse) | 0 | 1 | 1
  HL (PIF) | 0 | 2 | 2
Time between diagnosis to HCT [Count of Participants; unit: Participants]
  < 6 months | 14 | 10 | 24
  ≥ 6 months | 26 | 30 | 56
Number of prior autoHCTs [Count of Participants; unit: Participants]
  0 | 38 | 37 | 75
  1 | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Death from any cause. The time to this event is the time from HCT to death, loss to follow-up, or end of study (whichever comes first).
  The overall survival probability and 90% CI will be calculated by the Kaplan Meier product limit estimator.
Time Frame: 365 days post transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants | 72.3 [59.9 to 83.1] | 78.9 [66.9 to 88.8]

2. Secondary Outcome: Progression-free Survival
Description: Time from HCT until the documentation of disease progression / relapse or death due to any cause, whichever occurs first. Progression-free survival probability and 90% CI will be calculated by the Kaplan Meier product limit estimator.
Time Frame: 180 days and 365 days post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants
  180 days | 69.9 [57.4 to 81.1] | 72.5 [60.3 to 83.2]
  365 days | 62.1 [49.2 to 74.3] | 67.5 [54.9 to 79]

3. Secondary Outcome: Transplant-related Mortality
Description: Death without evidence of disease progression or recurrence. A cumulative incidence will be computed along with a 90% CI.
Time Frame: 100 days, 180 days, and 365 days post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants
  100 days | 5 [0.9 to 12.2] | 7.5 [2.1 to 15.8]
  180 days | 7.5 [2.1 to 15.8] | 7.5 [2.1 to 15.8]
  365 days | 7.5 [2.1 to 15.8] | 10 [3.6 to 19.2]

4. Secondary Outcome: Cumulative Incidence of Neutrophil Recovery
Description: Achieving a donor derived ANC ≥ 500/mm3 for 3 consecutive laboratory values on different days. A cumulative incidence will be computed along with a 90% CI.
Time Frame: 100 days and 365 days post transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants
  100 days | 97.5 [89.7 to 100] | 97.5 [89.8 to 100]
  365 days | 97.5 [89.7 to 100] | 97.5 [89.7 to 100]

5. Secondary Outcome: Cumulative Incidence of Platelet Recovery
Description: Achieving a platelet count ≥ 20,000/μL for 3 consecutive laboratory values on different days (with no platelet transfusions in the preceding seven days). A cumulative incidence will be computed along with a 90% CI.
Time Frame: 100 days and 365 days post transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants
  100 days | 87.5 [77 to 95.1] | 95 [86.2 to 99.5]
  365 days | 90 [79.7 to 96.9] | 95 [86.2 to 99.5]

6. Secondary Outcome: Cumulative Incidence of Acute GVHD
Description: Any skin, gastrointestinal or liver abnormalities fulfilling the BMT CTN Manual of Operations (2013) criteria of grades II-IV acute GVHD. A cumulative incidence will be computed along with a 90% CI.
  Any skin, gastrointestinal or liver abnormalities fulfilling the BMT CTN Manual of Operations (2013) criteria of grades III-IV acute GVHD. A cumulative incidence will be computed along with a 90% CI.
Time Frame: 100 days post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants
  Grades II-IV acute GVHD | 42.5 [29.8 to 55.7] | 32.5 [20.9 to 45.3]
  Grades III-IV acute GVHD | 17.5 [8.7 to 28.5] | 0 [0 to 0]

7. Secondary Outcome: Grades II-IV Acute GVHD
Description: Any skin, gastrointestinal or liver abnormalities fulfilling the BMT CTN Manual of Operations (2013) criteria of grades II-IV acute GVHD. A cumulative incidence will be computed along with a 90% CI.
Time Frame: 100 days
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants | 42.5 [29.8 to 55.7] | 32.5 [20.9 to 45.3]

8. Secondary Outcome: Grades III-IV Acute GVHD
Description: Any skin, gastrointestinal or liver abnormalities fulfilling the BMT CTN Manual of Operations (2013) criteria of grades III-IV acute GVHD. A cumulative incidence will be computed along with a 90% CI.
Time Frame: 100 days
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants | 17.5 [8.7 to 28.5] | 0 [0 to 0]

9. Secondary Outcome: Cumulative Incidence of Chronic GVHD
Description: Per National Institutes of Health (NIH) Consensus Criteria and includes organ involvement and severity, and overall global composite score (mild/moderate/severe). A cumulative incidence will be computed along with a 90% CI. Death from any cause. The time to this event is the time from HCT to death, loss to follow-up, or end of study (whichever comes first).
  The overall survival probability and 90% CI will be calculated by the Kaplan Meier product limit estimator.
Time Frame: 180 days and 365 days post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants
  180 days | 27.6 [16.7 to 40.2] | 10 [3.6 to 19.2]
  365 days | 35.5 [23.3 to 48.7] | 17.5 [8.7 to 28.5]

10. Secondary Outcome: Cumulative Incidences of Viral Reactivations and Infections: Grade 2-3 CMV Reactivation or Infection
Description: Grade 2: Clinically active CMV infection (e.g. symptoms, cytopenias) or CMV Viremia not decreasing by at least 2/3 of the baseline value after 2 weeks of therapy; Grade 3: CMV end-organ involvement (pneumonitis, enteritis, retinitis). A cumulative incidence will be computed along with a 90% CI. Death from any cause. The time to this event is the time from HCT to death, loss to follow-up, or end of study (whichever comes first).
  The overall survival probability and 90% CI will be calculated by the Kaplan Meier product limit estimator.
Time Frame: 100 days, 180 days, and 365 days
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants
  100 days | 10.4 [3.8 to 19.8] | 7.6 [2.2 to 16]
  180 days | 10.4 [3.8 to 19.8] | 7.6 [2.2 to 16]
  365 days | 10.4 [3.8 to 19.8] | 7.6 [2.2 to 16]

11. Secondary Outcome: Cumulative Incidences of Viral Reactivations and Infections: Grade 3 CMV Infection
Description: CMV end-organ involvement (pneumonitis, enteritis, retinitis) ). A cumulative incidence will be computed along with a 90% CI. Death from any cause. The time to this event is the time from HCT to death, loss to follow-up, or end of study (whichever comes first). The overall survival probability and 90% CI will be calculated by the Kaplan Meier product limit estimator.
Time Frame: 100 days, 180 days, and 365 days
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants
  100 days | 0 [0 to 0] | 2.6 [0.1 to 8.5]
  180 days | 0 [0 to 0] | 2.6 [0.1 to 8.5]
  365 days | 0 [0 to 0] | 2.6 [0.1 to 8.5]

12. Secondary Outcome: Cumulative Incidences of Viral Reactivations and Infections: Grade 2-3 EBV Infection
Description: Grade 2: EBV reactivation requiring institution of therapy with rituximab; Grade 3: EBV post-transplant lymphoproliferative disorder). A cumulative incidence will be computed along with a 90% CI. Death from any cause. The time to this event is the time from HCT to death, loss to follow-up, or end of study (whichever comes first). The overall survival probability and 90% CI will be calculated by the Kaplan Meier product limit estimator.
Time Frame: 100 days, 180 days, and 365 days
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants
  100 days | 0 [0 to 0] | 0 [0 to 0]
  180 days | 2.9 [0.1 to 9.5] | 0 [0 to 0]
  365 days | 2.9 [0.1 to 9.5] | 0 [0 to 0]

13. Secondary Outcome: Cumulative Incidences of Viral Reactivations and Infections: Grade 2 BK Virus Infection
Description: BK viremia or viruria with clinical consequence requiring prolonged therapy and/or surgical intervention). A cumulative incidence will be computed along with a 90% CI.
Time Frame: 100 days, 180 days, 365 days
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 38 | 37
percentage of participants
  100 days | 26.7 [15.7 to 39.2] | 29.7 [18.3 to 42.7]
  180 days | 26.7 [15.7 to 39.2] | 29.7 [18.3 to 42.7]
  365 days | 26.7 [15.7 to 39.2] | 29.7 [18.3 to 42.7]

14. Secondary Outcome: Cumulative Incidences of Viral Reactivations and Infections: Grade 2-3 Adenovirus Infection
Description: Grade 2: Adenoviral URI, viremia, or symptomatic viruria requiring treatment; Grade 3: ADV with end-organ involvement (except conjunctivitis and upper respiratory tract) ). A cumulative incidence will be computed along with a 90% CI. Death from any cause. The time to this event is the time from HCT to death, loss to follow-up, or end of study (whichever comes first). The overall survival probability and 90% CI will be calculated by the Kaplan Meier product limit estimator.
Time Frame: 100 days, 180 days, and 365 days
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 39 | 36
percentage of participants
  100 days | 2.6 [0.1 to 8.5] | 0 [0 to 0]
  180 days | 9 [2.6 to 18.9] | 9.4 [2.7 to 19.4]
  365 days | 9 [2.6 to 18.9] | 12.6 [4.6 to 23.8]

15. Secondary Outcome: Cumulative Incidences of Viral Reactivations and Infections: Grade 2 HHV-6 Infection
Description: Clinically active HHV-6 infection (e.g. symptoms, cytopenias) or HHV-6 viremia without viral load decline 0.5 log after 2 weeks of therapy). A cumulative incidence will be computed along with a 90% CI.
Time Frame: 100 days, 180 days, 365 days
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 39
percentage of participants
  100 days | 12.5 [5.3 to 22.3] | 5.1 [0.9 to 12.4]
  180 days | 12.5 [5.3 to 22.3] | 5.1 [0.9 to 12.4]
  365 days | 12.5 [5.3 to 22.3] | 5.1 [0.9 to 12.4]

16. Secondary Outcome: Cumulative Incidence of Relapse/Progression
Description: Defined by either morphological, cytogenetic/molecular or radiological evidence of disease consistent with pre-HCT features. A cumulative incidence will be computed along with a 90% CI. Death from any cause. The time to this event is the time from HCT to death, loss to follow-up, or end of study (whichever comes first). The overall survival probability and 90% CI will be calculated by the Kaplan Meier product limit estimator.
Time Frame: 180 days and 365 days post-transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants
  180 days | 22.6 [12.6 to 34.5] | 20 [10.6 to 31.5]
  365 days | 30.4 [18.9 to 43.2] | 22.5 [12.6 to 34.3]

17. Secondary Outcome: Cumulative Incidences of Thrombotic Microangiopathy (TMA) and Hepatic Veno-occlusive Disease (VOD)/Sinusoidal Obstruction Syndrome (SOS)
Description: TMA is defined as (Ho et al., 2005):
  1. RBC fragmentation and >2 schistocytes per high-power field on peripheral smear
  2. Concurrent increased serum LDH above institutional baseline
  3. Concurrent renal and/or neurologic dysfunction without other explanation
  4. Negative direct and indirect Coombs test results A cumulative incidence will be computed along with a 90% CI.
  VOD/SOS is defined as: In the first 20 days after HCT, the presence of ≥2 of the following: 1. Bilirubin >2 mg/Dl, 2. Hepatomegaly or pain in right upper quadrant, 3. Weight gain (>2% basal weight).
  A cumulative incidence will be computed along with a 90% CI.
Time Frame: 365 days post transplant
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
percentage of participants
  Thrombotic microangiopathy (TMA) | 5 [0.9 to 12.2] | 0 [0 to 0]
  Hepatic veno-occlusive disease (VOD)/sinusoidal obstruction syndrome (SOS) | 10 [3.6 to 19.2] | 2.5 [0.1 to 8.2]

18. Secondary Outcome: Cumulative Incidence of Primary Graft Failure
Description: Lack of donor-derived neutrophil engraftment. The frequency of subjects experiencing primary graft failure by 56 days will be described.
Time Frame: 56 days post-transplant
Population: Primary graft failure Lack of donor-derived neutrophil engraftment. The frequency of subjects experiencing primary graft failure by 56 days will be described. Transplanted participants surviving a minimum of 14 days post HCT and have complete data for both event status and event date.
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 39 | 40
Participants | 0 | 3

19. Secondary Outcome: Donor Chimerism
Description: Peripheral blood chimerism (% of donor chimerism) in whole blood (unsorted). The degree of donor chimerism will be summarized using descriptive statistics.
Time Frame: 28 days, 56 days, 100 days, 180 days, and 365 days post-transplant
Measure: Median (Full Range); unit: percentage of donor chimerism
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 34 | 39
percentage of donor chimerism
  28 days | 100 [92 to 100] | 99.1 [0 to 100]
  56 days | 100 [64 to 100] | 100 [0 to 100]
  100 days | 100 [43 to 100] | 100 [0 to 100]
  180 days | 100 [54.2 to 100] | 100 [43.9 to 100]
  365 days | 100 [79.4 to 100] | 100 [83.2 to 100]

20. Secondary Outcome: Peripheral Blood Chimerism
Description: The frequency of subjects with Peripheral blood (unsorted) chimerism>95% at 56 days will be described.
Time Frame: 56 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 26 | 32
Participants | 24 | 27

21. Secondary Outcome: Proportion of Subjects Proceeding to Transplant
Description: The proportion of subjects proceeding to HCT after informed consent.
Time Frame: Pre-HCT
Population: Participants who signed informed consent.
Measure: Count of Participants; unit: Participants
Groups:
- Overall Number of Participants Analyzed: Participants who signed informed consent.
Arm/Group | Overall Number of Participants Analyzed
Number analyzed (Participants) | 94
Participants | 80

22. Secondary Outcome: Time From Search to Donor Identification
Description: Time from search to donor identification Time from preliminary search to formal donor activation.
Time Frame: Pre-HCT
Measure: Median (Full Range); unit: days
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
days | 77.5 [16 to 733] | 88.5 [30 to 763]

23. Secondary Outcome: Donor Selection Characteristics: HLA Match
Description: Number of matched donor and recipient HLA allele pairs. A matched donor would have 8/8 HLA allele pairs matching; mismatched donors listed below have one to four mismatched HLA allele pairs at HLA-A, -B, -C, or -DRB1.
Time Frame: Pre-HCT
Measure: Count of Participants; unit: Participants
Groups:
- Total: Total number of participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC) | Total
Number analyzed (Participants) | 40 | 40 | 80
Participants
  7 out of 8 matching HLA allele pairs | 26 | 23 | 49
  6 out of 8 matching HLA allele pairs | 8 | 11 | 19
  5 out of 8 matching HLA allele pairs | 5 | 2 | 7
  4 out of 8 matching HLA allele pairs | 1 | 4 | 5

24. Secondary Outcome: Donor Selection Characteristics: Donor Age
Description: Donor age
Time Frame: Pre-HCT
Measure: Median (Full Range); unit: years
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC) | Total
Number analyzed (Participants) | 40 | 40 | 80
years | 27 [18 to 56] | 29 [21 to 44] | 29 [18 to 56]

25. Secondary Outcome: Donor Selection Characteristics: Donor Age, Categorical
Description: Donor age, categorical
Time Frame: Pre-HCT
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC) | Total
Number analyzed (Participants) | 40 | 40 | 80
Participants
  18-29 | 24 | 23 | 47
  30-39 | 9 | 11 | 20
  40-49 | 4 | 6 | 10
  50-59 | 3 | 0 | 3

26. Secondary Outcome: Donor Selection Characteristics: Donor Weight
Description: Donor weight
Time Frame: Pre-HCT
Measure: Median (Full Range); unit: kg
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC) | Total
Number analyzed (Participants) | 40 | 40 | 80
kg | 77 [55 to 103] | 77 [52 to 104] | 77 [52 to 104]

27. Secondary Outcome: Donor Selection Characteristics: Donor Sex
Description: Donor sex
Time Frame: Pre-HCT
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC) | Total
Number analyzed (Participants) | 40 | 40 | 80
Participants
  Male | 20 | 24 | 44
  Female | 20 | 16 | 36

28. Secondary Outcome: Donor Selection Characteristics: Donor and Recipient Sex
Description: Donor-recipient sex match
Time Frame: Pre-HCT
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC) | Total
Number analyzed (Participants) | 40 | 40 | 80
Participants
  Male and male | 12 | 12 | 24
  Male and female | 8 | 12 | 20
  Female and male | 11 | 7 | 18
  Female and female | 9 | 9 | 18

29. Secondary Outcome: Donor Selection Characteristics: Donor and Recipient CMV Serostatus
Description: Donor-recipient Cytomegalovirus (CMV) serostatus match
Time Frame: Pre-HCT
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC) | Total
Number analyzed (Participants) | 40 | 40 | 80
Participants
  +/+ | 18 | 13 | 31
  +/- | 6 | 5 | 11
  -/+ | 9 | 10 | 19
  -/- | 7 | 12 | 19

30. Secondary Outcome: Donor Selection Characteristics: Donor and Recipient ABO Blood Match
Description: Donor-recipient ABO group match
Time Frame: Pre-HCT
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC) | Total
Number analyzed (Participants) | 40 | 40 | 80
Participants
  Matched | 20 | 24 | 44
  Minor mismatch | 12 | 5 | 17
  Major mismatch | 8 | 8 | 16
  Bidirectional | 0 | 3 | 3

31. Secondary Outcome: Donor Clonal Hematopoiesis
Description: The proportion of subjects developing donor clonal hematopoiesis
Time Frame: 100 days and 365 days post-transplant
Population: All participants assessed for donor clonal hematopoiesis.
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 40 | 40
Participants | 0 | 0

32. Secondary Outcome: Subgroup Analysis of HIV-positive Subjects
Description: If CCR5delta32 homozygous donors are successfully found and used for one or more HIV-positive subjects, a descriptive analysis of baseline characteristics and outcomes for those HIV-positive subjects will be conducted, including the viral load detected over time obtained from collected samples.
Time Frame: 365 days post transplant
Population: Four subjects with HIV-positive, no statistical analysis for this outcome measure was completed due to limited HIV-positive rate. Descriptive analysis provided.
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 0 | 4
Participants
  Survival Status: Alive | 0 | 1
  Survival Status: Deceased (relapse) | 0 | 2
  Survival Status: Deceased (fungal infection) | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 1 year post transplant
Description: Evaluation of toxicities will be graded using National Cancer Institute Common Toxicity Criteria, specifically CTCAE version 4.03. The protocol pre-specifies that Adverse Events on this study are reported and evaluated by conditioning regimen arm (MAC or RIC).
Arm/Group | Myeloablative Conditioning (MAC) | Reduced Intensity Conditioning (RIC)
All-Cause Mortality (participants affected / at risk) | 11/40 | 8/40
Serious Adverse Events (participants affected / at risk) | 12/40 | 13/40
Other Adverse Events (participants affected / at risk) | 5/40 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Myeloablative Conditioning (MAC) (N=40) | Reduced Intensity Conditioning (RIC) (N=40)
Other (Blood and lymphatic system disorders) | 2 | 0 — Recurrence, persistence, or progression of disease
Other (Eye disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 2
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 3
Sinusitis (Infections and infestations) | 0 | 1
Other (Infections and infestations) | 1 | 0
Other (Investigations) | 1 | 0
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 — One case of Acute Myeloid Leukemia under MAC, two cases of recurrence, persistence, or progression of disease under MAC, and two cases of recurrence, persistence, or progression of disease under RIC.
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Myeloablative Conditioning (MAC) (N=40) | Reduced Intensity Conditioning (RIC) (N=40)
Myocardial infarction (Cardiac disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT02793544/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-16): https://cdn.clinicaltrials.gov/large-docs/44/NCT02793544/ICF_001.pdf